CLINICAL TRIAL: NCT03433599
Title: Repetitive Acute Intermittent Hypoxia for Spinal Cord Repair
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Shirley Ryan AbilityLab (Other)
Collaborators: U.S. Department of Education (U.S. Federal Agency)
Responsible Party: Principal Investigator, Monica Perez, Scientific Chair Arms + Hands AbilityLab, Shirley Ryan AbilityLab
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: STU00212000
Record Dates: First submitted 2018-02-08; First posted 2018-02-14 (Actual); Last update posted 2022-06-30 (Actual); Status verified 2022-06

CONDITIONS: Spinal Cord Injuries
Keywords: Acute Intermittent Hypoxia; Transcranial Magnetic Stimulation
MeSH Terms: conditions — Spinal Cord Injuries

STUDY DESIGN:
Who Masked: Participant, Care Provider
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- rAIH + training by research staff (Active Comparator): Participants will receive repeated exposure to acute Intermittent Hypoxia (rAIH) and training by research staff.
  Interventions: Other: Repeated exposure to acute Intermittent Hypoxia (rAIH); Other: Upper-limb Training by Research Staff; Other: Lower-limb Training by Research Staff
- sham rAIH + training (Sham Comparator): Participants will sham receive repeated exposure to acute Intermittent Hypoxia (rAIH) and training by the research staff.
  Interventions: Other: Normal Room Air; Other: Upper-limb Training by Research Staff; Other: Lower-limb Training by Research Staff

INTERVENTIONS:
Other: Repeated exposure to acute Intermittent Hypoxia (rAIH) — Participants will be fitted with a mask that will be placed over mouth and nose. Tubing will be attached to the front of the mask. The session will last approximately 30-45 minutes with 60-90 seconds of lower oxygen (tubing attached, 9-10% oxygen level), alternating with 60-90 sec of normal room air (no tubing attached).
  Arms: rAIH + training by research staff
Other: Normal Room Air — Participants will be fitted with a mask that will be placed over mouth and nose. Tubing will be attached to the front of the mask. The session will last approximately 30-45 minutes with 60-90 seconds of normal room air (with tubing attached to the mask) and 60-90 sec of normal room air (without the tubing attached to the mask).
  Other Names: Sham repeated exposure to acute Intermittent Hypoxia (rAIH)
  Arms: sham rAIH + training
Other: Upper-limb Training by Research Staff — Training sessions will last for approximately 30 minutes, with additional time for set up. During these sessions, participants will be asked to complete a variety of tasks related to general arm/hand movement, gross grasping, fine grasping, and hand cycle using an arm ergometer. The number of repetitions will be monitored and adjust the difficulty to ensure appropriate task difficulty.
Other: Lower-limb Training by Research Staff — Training sessions will last for approximately 30 minutes, with additional time for set up. During these sessions, participants will be asked to complete a variety of tasks related to general leg/foot movement, over-ground walking, treadmill walking, stair climbing training, leg cycling, standing frame, and NuStep. The number of repetitions will be monitored and adjust the difficulty to ensure appropriate task difficulty.

SUMMARY:
Our goal is to enhance repeated exposure to acute intermittent hypoxia (rAIH)/training-induced aftereffects on upper and lower limb function recovery in humans with chronic spinal cord injury (SCI).

DETAILED DESCRIPTION:
The experiments in this study will test the following: Hypothesis 1.1(Experiment 1) that rAIH will enhance corticospinal excitability and upper and lower limb function in humans with incomplete SCI. Hypothesis 1.2 (Experiment 2) that enhancing the aftereffects of rAIH with exercise training will further enhance upper and lower limb motor function in humans with incomplete SCI. Measurements of corticospinal, cortical, and motoneuron excitability will be tested to further understand the mechanisms of this induced-plasticity. Persons with chronic (>6 months) spinal cord injury between the levels of C2 and T2. SCI subjects must possess either the ability to produce a visible precision grip force with one hand, and/or the ability to perform some small wrist flexion and extension. Additionally, subject must possess the ability to perform a small visible contraction with dorsiflexion and hip flexor muscles. Controls must be right handed due to potential differences in the organization of the brain in right handed and left handed individuals.

ELIGIBILITY:
Inclusion criteria for SCI:

1. Males and females between 18-85 years
2. Chronic SCI (≥ 6 months post injury)
3. SCI at or above L2
4. ASIA A, B, C, or D, complete or incomplete
5. Possess the following: The ability to produce a visible precision grip force with one hand, and/or the ability to perform some small wrist flexion and extension. The ability to perform a small visible contraction with dorsiflexion and hip flexor muscles.

Inclusion criteria for controls:

1. Males and females between 18-85 years
2. Right-handed (Only right-handed individuals will be accepted into this group because of the potential differences in the organization of the brain in right handed and left handed individuals)

Exclusion criteria for SCI and for controls:

1. Uncontrolled medical problems including pulmonary, cardiovascular or orthopedic disease
2. Any debilitating disease prior to the SCI that caused exercise intolerance
3. Premorbid, ongoing major depression or psychosis, altered cognitive status
4. History of head injury or stroke
5. Metal plate in skull
6. History of seizures
7. Receiving drugs acting primarily on the central nervous system, which lower the seizure threshold such as antipsychotic drugs (chlorpromazine, clozapine) or tricyclic antidepressant
8. Pregnant females
9. Ongoing cord compression or a syrinx in the spinal cord or a spinal cord disease as spinal stenosis, spina bifida or herniated cervical disk.

AIH exclusion criteria (in addition to the above listed exclusion criteria)

1. Resting heart rate ≥120 BPM
2. Resting systolic blood pressure >180 mm Hg
3. Resting diastolic Blood Pressure >100 mmHg
4. Self-reported history of unstable angina or myocardial infarction within the previous month
5. Resting SpO2 ≥ 95%
6. Cardiopulmonary complications such as COPD

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2020-04-09 (Actual); Primary Completion 2024-12-28 (Estimated); Study Completion 2025-12-28 (Estimated)

PRIMARY OUTCOMES:
Upper limb functional measurement | 45 minutes to 1 hour
  The Graded Redefined Assessment of Strength, Sensibility and Prehension (GRASSP) will be used to assess sensation, strength, and prehension.
Lower limb functional measurement | 5-10 minutes
  10-meter walk test will be used to assess walking speed
MEP/CMEP recruitment curves using TMS | 30 minutes to 1 hour
  Ten Transcranial magnetic stimuli (TMS) will be delivered to plot the mean peak-to-peak amplitude of the motor and cervicomedullary evoked potentials (MEPs and CMEPs, respectively) from the non-rectified response against the TMS intensity in each subject (MEP/CMEP recruitment curves).
EMG and force voluntary output | 30 minutes to 1 hour
  EMG surface electrodes will be placed over target muscles (deltoid, biceps brachii, first dorsal interosseous, abductor pollicis brevis, quadriceps femoris, tibialis anterior and/or soleus) to measure maximum voluntary contraction (MVC)

CONTACTS AND LOCATIONS:
Overall Officials: Monica A Perez, PhD, Principal Investigator — Shirley Ryan AbilityLab
Locations (1):
- Shirley Ryan AbilityLab, Chicago, Illinois, United States